CLINICAL TRIAL: NCT03216707
Title: The Effects of High Definition Transcranial Direct Current Stimulation Over Primary Motor Cortex Versus Insular Cortical Targets on Experimental Capsaicin Induced Hyperalgesia and Pain in Healthy Volunteers
Brief Title: High Definition Transcranial Direct Current Stimulation Motor Cortex Versus Insula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Collaborators: Swansea University (Other); University College London Hospitals (Other)
Responsible Party: Principal Investigator, Saeid Metwaly Abouelyazid Elsawy, Principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RSO
Record Dates: First submitted 2017-07-06; First posted 2017-07-13 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- HD tDCS sham motor cortex (Sham Comparator): the intervention 10 participants will be subjected to1.5 gram of Capsaicin cream 0.075% concentration for 30 min then participants will be subjected to sham stimulation targeting motor cortex area using the high-definition transcranial direct current stimulation device by starting stimulation for 30 seconds then stop stimulation for 20 min
  Interventions: Device: HD tDCS sham motor cortex; Other: Capsaicin cream
- HD tDCS active motor cortex (Active Comparator): the intervention will be 10 participants will be subjected to 1.5-gram of Capsaicin cream 0.075 concentration for 30 min then participants will be subjected to active stimulation targeting motor cortex area with the high-definition transcranial direct current stimulation device with current intensity 2 milliampere for 20 min
  Interventions: Device: HD tDCS active motor cortex; Other: Capsaicin cream
- HD tDCS active insula cortex (Active Comparator): the intervention will be 10 participants will be subjected to 1.5 gram of Capsaicin cream 0.075 concentration for 30 min then participants will be subjected to active stimulation targeting Insular cortex area with the high-definition transcranial direct current stimulation device, with current intensity 2milliampere for 20 min
  Interventions: Device: HD tDCS active insula cortex; Other: Capsaicin cream

INTERVENTIONS:
Device: HD tDCS active motor cortex — the intervention will be 10 participants will be subjected to 1.5-gram of Capsaicin cream 0.075 concentration for 30 min then participants will be subjected to active stimulation targeting motor cortex area with the high-definition transcranial direct current stimulation device with current intensity 2 milliampere for 20 min
  Arms: HD tDCS active motor cortex
Device: HD tDCS active insula cortex — the intervention will be 10 participants will be subjected to 1.5 gram of Capsaicin cream 0.075 concentration for 30 min then participants will be subjected to active stimulation targeting Insular cortex area with the high-definition transcranial direct current stimulation device, with current intensity 2milliampere for 20 min
  Arms: HD tDCS active insula cortex
Device: HD tDCS sham motor cortex — the intervention 10 participants will be subjected to1.5 gram of Capsaicin cream 0.075% concentration for 30 min then participants will be subjected to sham stimulation targeting motor cortex area using the high-definition transcranial direct current stimulation device by starting stimulation for 30 seconds then stop stimulation for 20 min
  Arms: HD tDCS sham motor cortex
Other: Capsaicin cream — Capsaicin cream

SUMMARY:
Brain stimulation is a technique that can alter cortical function and thus be suitable for treating pain. This is especially when pain is chronic and associated with functional and even structural reorganization of the central nervous system. The idea of using invasive and noninvasive brain stimulation for pain relief is not new. Studies from the 1950s have investigated the brain stimulation for therapeutic use. Direct implantation of electrodes on the cerebral cortex has been carried out by Tsubokawa and colleagues in Japan. Although reported to be effective, it is invasive and involves the implantation of a foreign body into the cranium. Recent advancements in the techniques of non-invasive brain stimulation have improved and have measurable modulatory effects making this an attractive alternative for treating pain

DETAILED DESCRIPTION:
Repetitive transcranial magnetic stimulation and transcranial direct current stimulation are currently the two main methods of non-invasive brain stimulation under investigation. Stimulation of the primary motor cortex has been reported to relieve neuropathic, musculoskeletal, visceral pain as well as headaches and migraine. Other parameters of stimulation have shown encouraging results. For example, stimulation of the secondary somatosensory cortex was also reported to relieve chronic visceral pain. However, there are numerous unanswered questions regarding these techniques.

This research project is an attempt to answer some of these questions:

1. Which pain conditions can be alleviated by non-invasive brain stimulation?
2. What are the best parameters for stimulation-

   1. method: transcranial direct current stimulation or repetitive transcranial magnetic stimulation transcranial or Alternating Current Stimulation
   2. High-Definition transcranial direct current stimulation or conventional transcranial direct current stimulation?
   3. which area to stimulate? Primary motor cortex, insula?
3. Will other forms of treatment such as pharmacotherapy, peripheral nerve stimulation or multi-disciplinary pain management enhance the effectiveness of non-invasive brain stimulation

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent to participate in the study.
* Male and female University Undergraduate, Postgraduate and staff in the Department of Psychology.
* American society of anesthesiology scores I to II patients.

Exclusion Criteria: the participant who has any history of:

* an adverse reaction to brain stimulation.
* a seizure
* an unexplained loss of consciousness
* a stroke
* serious head injury
* surgery to their head
* any brain related, neurological illnesses
* any illness that may have caused brain injury
* frequent or severe headaches
* metal in your head (outside the mouth) such as shrapnel, surgical clips, or fragments from welding
* any implanted medical devices such as cardiac pacemaker's or medical pumps
* taking any analgesic medications in the past 24 hours
* pregnancy
* anyone in your family has epilepsy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Pain severity assessment using Numerical Rating Scale (NRS score from 0-100) | 30 min after capsaicin cream application and at the end of the HD tDCS session and one hour after study
  we will put the capsaicin cream for 30 min at an area of 9 cm2 then we will assess the pain score throughout this time of application of the cream every 5 min

SECONDARY OUTCOMES:
map area of sensitization caused by application of capsaicin cream | 30 min after the capsaicin cream application and at the end of HD tDCS sessionand one hour after study
  The area of sensitization using calibrated Neurotip test using the spring mechanism which will exert a force of 40 gm so we will detect the change in sensation to the pin brick in the area of cream application

CONTACTS AND LOCATIONS:
Locations (1):
- Saeid Elsawy, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided